CLINICAL TRIAL: NCT00000983
Title: A Randomized Blinded Trial To Evaluate the Safety and Tolerance of High Versus Low Dose Zidovudine Administered to Children With Human Immunodeficiency Virus
Brief Title: The Safety of Different Dose Levels of Zidovudine in HIV-Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 128; 11103 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate and compare differences in tolerance and side effects associated with two different dosages of zidovudine (AZT) when used to treat children with HIV infection. Other goals are to evaluate and compare the degree of change in neurodevelopmental disease and determine whether there are differences in the rate and degree of toxicities associated with one versus the other dosage.

AZT has been shown to decrease the death rate and frequency of opportunistic infections in certain adult patients with symptomatic HIV infection. Thus, it is likely that symptomatic HIV infected children may also benefit from AZT. Studies of the safety and pharmacokinetics (blood levels) in children have indicated that AZT can be given to children in doses that can be tolerated and that can be assumed to be therapeutic. Those currently taking care of infected children no longer feel it is ethical to conduct an AZT/placebo (inactive substance) trial. In addition, given the information learned from studies of adult patients that shows effectiveness of AZT at lower doses, experience with an equivalent lower dose in children needs to be studied.

DETAILED DESCRIPTION:
AZT has been shown to decrease the death rate and frequency of opportunistic infections in certain adult patients with symptomatic HIV infection. Thus, it is likely that symptomatic HIV infected children may also benefit from AZT. Studies of the safety and pharmacokinetics (blood levels) in children have indicated that AZT can be given to children in doses that can be tolerated and that can be assumed to be therapeutic. Those currently taking care of infected children no longer feel it is ethical to conduct an AZT/placebo (inactive substance) trial. In addition, given the information learned from studies of adult patients that shows effectiveness of AZT at lower doses, experience with an equivalent lower dose in children needs to be studied.

All participants are randomized to receive AZT at 1 of 2 doses. Patients are stratified according to whether CD4 cell counts are > or < 500 cells/mm3 as well as whether symptoms are mild to moderate or if patients have lymphocytic interstitial pneumonitis (LIP). Medication is dispensed every other week for the first 8 weeks and monthly until week 104, then either monthly or every 3 months. Safety and effectiveness of the treatment program are evaluated at 6-month intervals to assess whether it is appropriate to continue the study as originally designed. Patients are evaluated every 2 weeks for the first 8 weeks, monthly until week 104, every 3 months until week 208, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

AMENDED:

* 03-19-91 Prophylaxis for PCP is recommended according to current practice guidelines. As per published recommendations, primary prophylaxis with TMP / SMX on a M-T-W basis is encouraged.

Allowed:

* Immunoglobulin therapy as single dose exposure prophylaxis or for children with hypogammaglobulinemia.
* Trimethoprim / sulfamethoxazole (TMP / SMX) and parenteral or aerosolized pentamidine for prophylaxis for Pneumocystis carinii pneumonia for children with AIDS and/or CD4+ counts = or < 500 cells/mm3.
* Systemic ketoconazole and acyclovir, or oral nystatin for acute therapy.
* Aerosol ribavirin for short-term treatment of acute respiratory syncytial virus (RSV).

AMENDED:

* 9/17/90 enrollment is limited to children < 6 years of age.
* Original design:
* Patients must have the following:
* Parent or guardian available to give written informed consent.
* Laboratory evidence of HIV infection.
* Children < 15 months of age, with CD4+ cell count > 500 cells/mm3, who are thought to have acquired HIV through perinatal transmission and whose only laboratory evidence of HIV infection is a positive antibody test, must also have one or more of the laboratory criteria described in Disease Status AND one or more of the disease criteria that are required of children > 15 months old with CD4+ cell counts > 500 cells/mm3.

Prior Medication:

Allowed:

* Aerosol ribavirin.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

Previous AIDS-defining opportunistic infection or neoplasms as specified by the CDC surveillance criteria for AIDS.

* Previous unexplained recurrent, serious bacterial infections (two or more within a 2-year period) including sepsis, meningitis, pneumonia, abscess of an internal organ, and bone/joint infections caused by Haemophilus, Streptococcus, or other pyogenic bacteria.
* Qualifying for entrance criteria to zidovudine (AZT) + or - gammaglobulin (ACTG 051).
* Encephalopathy.
* Failure to thrive (defined as a child who crosses two percentile lines on the growth chart or child who is < fifth percentile and does not follow curve) and/or oral candidiasis for at least 2 months despite appropriate topical therapy.
* Lymphocytic interstitial pneumonitis (LIP) with steroid dependency or requiring supplemental oxygen.
* Preexisting malignancies.

Concurrent Medication:

AMENDED:

* 03-19-91 Prophylaxis with antiviral or antifungals agents, except for PCP prophylaxis is prohibited.
* Drugs that are metabolized by hepatic glucuronidation should be used with caution.

Excluded:

* Prophylaxis for oral candidiasis or otitis media or other infections (sinusitis, urinary tract infections).
* Immunoglobulin therapy not specifically allowed.
* Ketoconazole, acyclovir, or nystatin for prophylaxis.
* Drugs that are metabolized by hepatic glucuronidation and might alter metabolism of zidovudine (AZT).

Patients with the following are excluded:

* Previous AIDS-defining opportunistic infection or neoplasms as specified by the CDC surveillance criteria for AIDS.
* Previous unexplained recurrent, serious bacterial infections (two or more within a 2-year period) including sepsis, meningitis, pneumonia, abscess of an internal organ, and bone/joint infections caused by Haemophilus, Streptococcus, or other pyogenic bacteria.
* Qualifying for entrance criteria to zidovudine (AZT) + or - gammaglobulin (ACTG 051).
* Encephalopathy.
* Failure to thrive (defined as a child who crosses two percentile lines on the growth chart or child who is < fifth percentile and does not follow curve) and/or oral candidiasis for at least 2 months despite appropriate topical therapy.
* Lymphocytic interstitial pneumonitis (LIP) with steroid dependency or requiring supplemental oxygen.
* Preexisting malignancies.

Prior Medication:

Excluded within 2 weeks of study entry:

* Any other experimental therapy or drugs that cause prolonged neutropenia or significant nephrotoxicity.

Excluded within 1 month of study entry:

* Antiretroviral agents.
* Immunomodulating agents including immunoglobulin, interferon, isoprinosine, and IL-2.

Excluded within 2 months of study entry:

* Systemic ribavirin for retroviral therapy.

Prior Treatment:

Excluded within 1 month of study entry:

* Lymphocyte or red blood cell transfusions.

Active alcohol or drug abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Study Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Brady, Study Chair; P Weintrub, Study Chair
Locations (51):
- United States (48):
  - Kaiser Permanente / UCLA Med Ctr, Downey, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Northern California Pediatric AIDS Treatment Ctr / UCSF, San Francisco, California
  - Univ of Connecticut Health Ctr / Pediatrics, Farmington, Connecticut
  - Children's Natl Med Ctr, Washington D.C., District of Columbia
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - SUNY / Health Sciences Ctr at Brooklyn / Pediatrics, Brooklyn, New York
  - Jewish Hosp Ctr of Long Island / Pediatrics, Jamaica, New York
  - Schneider Children's Hosp / Long Island Jewish Med Ctr, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Univ Babies' Hosp, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Lincoln Hosp Ctr / Pediatrics, The Bronx, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Westchester Hosp / New York Med College / Pediatrics, Valhalla, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - San Juan City Hosp, San Juan
  - UPR Children's Hosp / San Juan City Hosp, San Juan

REFERENCES:
- [Background] Lathey JL, Marschner IC, Kabat B, Spector SA. Deterioration of detectable human immunodeficiency virus serum p24 antigen in samples stored for batch testing. J Clin Microbiol. 1997 Mar;35(3):631-5. doi: 10.1128/jcm.35.3.631-635.1997. PMID 9041402
- [Background] Fiscus SA, Welles SL, Spector SA, Lathey JL. Length of incubation time for human immunodeficiency virus cultures. J Clin Microbiol. 1995 Jan;33(1):246-7. doi: 10.1128/jcm.33.1.246-247.1995. PMID 7699053
- [Background] Brady MT, McGrath N, Brouwers P, Gelber R, Fowler MG, Yogev R, Hutton N, Bryson YJ, Mitchell CD, Fikrig S, Borkowsky W, Jimenez E, McSherry G, Rubinstein A, Wilfert CM, McIntosh K, Elkins MM, Weintrub PS. Randomized study of the tolerance and efficacy of high- versus low-dose zidovudine in human immunodeficiency virus-infected children with mild to moderate symptoms (AIDS Clinical Trials Group 128). Pediatric AIDS Clinical Trials Group. J Infect Dis. 1996 May;173(5):1097-106. doi: 10.1093/infdis/173.5.1097. PMID 8627060
- [Background] Brady M, McGrath N, Brouwers P, Gelber R, Fowler M, Weintrub P. Controlled trial of tolerance and efficacy of zidovudine (ZDV) at standard and low dose in children (ACTG 128). The Pediatric AIDS Clinical Trials Group. Int Conf AIDS. 1994 Aug 7-12;10(1):79 (abstract no 268B)
- [Background] Parent D, Ellner J, Hafner R, Williams M, Jacobs P, Hojczyk P. A phase II/III trial of Rifampin (RIF) Ciprofloxach (CIPRO), Clofazimine (CLOF), Ethambutol (ETH), +/- Amikacin (AK) in the treatment (RX) of Disseminated Mycobacterium avium (MA) infection in HIV-infected individuals (PTS). Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:56
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891